CLINICAL TRIAL: NCT00673413
Title: The Perception of the Estomy-Individual Regarding of Its Situation
Status: Completed | Type: Observational
Sponsor: Universidade da Regiao da Campanha (Other)
Collaborators: Secretary of Health and Environment Bagé (Unknown)
Responsible Party: Region of Campaign University, Center for Pharmaceutical Assistance
Other Study IDs: X12605
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Health Promotion; Health Behavior; Pharmaceutical Services; Psychology, Clinical
Keywords: Perception; Emotions; Adaptation; Estomia
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The present work had as purpose to analyze estomy-individuals according to the feelings of their current situation.

DETAILED DESCRIPTION:
The present work had as purpose to analyze estomy-individuals according to the feelings of their current situation. It is about a descriptive research of qualitative approach that took place in September, 2006. The population under study was composed by five estomy patients participants in a Grupo de Atenção dos Estomizados, which has multi-disciplinary character, at the Universidade da Região da Campanha (URCAMP) in the city of Bagé in South Brazil. The collection of data was given through not structuralized interviews and with the estomy-individuals, after the same ones read and signed the term of informed free ssent. The data form analyzed through the method of analysis of categories. Each one received a denomination with capital letters from the alphabet (A, B, D, and E) for their identification. The most significant categories in the answers from the ones being tested were manifestations and feelings of daptation, resignation and affective bond.The manifestation of anger and suffering shown by subjects D and E were only mentioned in this study, not being considered categories. The feeling shown by subjects A, B and C show an acceptance of their reality as rehabilitated from a surgical procedure, in the attempt of decreasing the psycho suffering caused by the mutilation and adaptation to the new status quo, fact which was observed for not appearing in the answers feeling such as revolt and guilty, which are mentioned in the review of literature as characteristics of subjects who suffered a surgical intervention. It is noticed that family support is a determinant fact to accept the new reality. The study contributed to know the subjectivity of the estomated, opening possibilities to improve the attention to health by the multi-professional staff.

Descriptors: Perception; emotions; Adaptation; estomia

ELIGIBILITY:
Inclusion Criteria:

* Estomizados registered in the Single Health System users group's support of the University.

Exclusion Criteria:

* Estomizados unable to come to the group of support for health reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Estomizados of a group of visitors to estomizados support from the Center for Pharmaceutical Assistance at the University of the Region Campaign.
Sampling Method: Non-Probability Sample
Dates: Start 2006-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade da Região da Campanha, Bagé, Rio Grande do Sul, Brazil